CLINICAL TRIAL: NCT04995627
Title: Exploratory Study Into the Effect of Salt Supplementation in Gitelman Syndrome
Brief Title: Salt Supplementation in Gitelman Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Kidney Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL72495.091.19
Record Dates: First submitted 2021-07-18; First posted 2021-08-09 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Gitelman Syndrome
MeSH Terms: conditions — Gitelman Syndrome | interventions — Salts

STUDY DESIGN:
Intervention Model Description: Single subject multiple randomized double-blinded multi-crossover placebo-controlled trials (N-of-1 trials)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salt (NaCl) (Active Comparator): 12 grams (12 capsules) of NaCl per day
  Note: participants will be treated with active and placebo comparator (N-of-1 trial design)
  Interventions: Dietary Supplement: Salt (NaCl)
- Placebo (Placebo Comparator): 12 capsules of placebo per day
  Note: participants will be treated with active and placebo comparator (N-of-1 trial design)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Salt (NaCl) — 12 grams of salt (NaCl) per day
  Arms: Salt (NaCl)
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of salt (NaCl) supplementation on serum potassium and clinical signs and symptoms in patients with Gitelman syndrome.

DETAILED DESCRIPTION:
Single subject multiple randomized double-blinded multi-crossover placebo-controlled trials (N-of-1 trials) will be performed. Participants will enroll the study after giving written informed consent. The individual trials will consist of 3 treatment blocks which each contain a 4-week treatment period of salt supplementation (12 grams of NaCl) and a 4-week treatment period of placebo, in a randomized, blinded order. After each period of 4 weeks, outcomes measures will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Genetically-proven, symptomatic Gitelman syndrome
* Written informed consent

Exclusion Criteria:

* inability to discontinue potassium-sparing diuretics, mineralocorticoid antagonists and NSAIDs; this means inability to reach a potassium level of 2.5 mmol/L or higher with maximally tolerable potassium supplementation after discontinuation of potassium-sparing diuretics
* pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in serum Potassium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum potassium
Change in symptoms measured by personalized symptom score sheet | Weekly (week 0 till week 24)
  Symptoms will be scored via a personalized symptom score sheet, which will be composed with the individual participant. Symptoms will be scored at a range from 0 - 10

SECONDARY OUTCOMES:
Change in serum sodium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum sodium
Change in serum magnesium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum magnesium
Change in serum chloride | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum chloride
Change in serum bicarbonate | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum bicarbonate
Change in serum calcium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum calcium
Change in serum creatinine | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum creatinine
Change in serum aldosterone | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum aldosterone
Change in serum renin | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in serum renin
Change in fractional urinary excretion of potassium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in fractional urinary excretion of potassium
Change in fractional urinary excretion of sodium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in fractional urinary excretion of sodium
Change in fractional urinary excretion of chloride | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in fractional urinary excretion of chloride
Change in fractional urinary excretion of magnesium | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in fractional urinary excretion of magnesium
Change in urinary calcium/creatinine ratio | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in urinary calcium/creatinine ratio
Change in urinary excretion of renin | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in urinary excretion of renin
Change in urinary excretion of aldosterone | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Change in urinary excretion of aldosterone
Gitelman symptom questionnaire | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  With the Gitelman symptom questionnaire, symptoms can be scored for frequency of apperance and severity. This questionnaire also contains the 36-Item Short Form Health Survey (RAND SF-36) quality of life questionnaire
Blood pressure (including orthostatic hypotension measurement) | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Measurement of blood pressure including measurement of orthostatic blood pressure
Weight | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Body Weight
Muscle strength | Baseline, week 4, week 8, week 12, week 16, week 20, week 24
  Muscle strength will be measured by hand grip dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Tom Nijenhuis, MD PhD, Principal Investigator — Radboud University Medical Center
Locations (3):
- University Hospital of University of Campania "L. Vanvitelli", Naples, Italy
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Erasmus MC, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: Undecided